CLINICAL TRIAL: NCT00486720
Title: A Randomized Phase IIa Study of Vorinostat in Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Phase IIa Vorinostat (MK0683, Suberoylanilide Hydroxamic Acid (SAHA)) Study in Lower Risk Myelodysplastic Syndromes (0683-064)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0683-064; MK0683-064; 2007_536
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Results first posted 2010-06-22 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: Myelodysplastic Syndromes; Blood Disease; Bone Marrow Disease
MeSH Terms: conditions — Myelodysplastic Syndromes; Hematologic Diseases; Bone Marrow Diseases | interventions — Vorinostat

ARMS (2):
- 1 (Experimental): vorinostat 400 mg
  Interventions: Drug: vorinostat
- 2 (Experimental): vorinostat 200 mg
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — vorinostat 400 mg by mouth (P.O.) capsules once daily (q.d.). Treatment in 21 day cycles for up to 8 cycles.
  Other Names: suberoylanilide hydroxamic acid (SAHA); ZOLINZA®
  Arms: 1
Drug: vorinostat — vorinostat 200 mg by mouth (P.O.) capsules three times daily (t.i.d.). Treatment in 21 day cycles for up to 8 cycles.
  Other Names: suberoylanilide hydroxamic acid (SAHA); ZOLINZA®
  Arms: 2

SUMMARY:
This study is to evaluate the efficacy, safety and tolerability of vorinostat in patients with lower risk Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

Patient is a male or female, at least 18 years of age with low or intermediate-1 risk Myelodysplastic Syndrome (MDS) defined by the International Prognostic Scoring System

* Patient has previously untreated disease, or has received up to one prior treatment regimen for lower-risk Myelodysplastic Syndrome
* Patient has a performance status of equal to or less than 2 on the Eastern Cooperative Oncology Group Performance Scale
* Patient must have adequate organ function

Exclusion Criteria:

* Patient has clinical evidence of Central Nervous System (CNS) leukemia
* Patient is pregnant or breastfeeding, or expecting to conceive within the projected duration of the study
* Patient had prior treatment with a histone deacetylase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first patient in was 26-Jun-2007. The date of last patient last visit for the study was 16-Jul-2009.
Pre-assignment Details: Vorinostat was studied in patients who were first stratified by their International Prognostic Scoring System
  for myelodysplastic syndrome (low versus intermediate-1) and than randomized into one of two dose schedules.
Groups:
- Vorinostat Once Daily Dose Schedule: Vorinostat 400 mg once daily for 14 consecutive days in a 21 day cycle.
- Vorinostat Thrice Daily Dose Schedule: Vorinostat 200 mg three times daily for 14 consecutive days in a 21 day cycle.
Period: Overall Study
Arm/Group | Vorinostat Once Daily Dose Schedule | Vorinostat Thrice Daily Dose Schedule
Started | 10 (1 randomized patient was discontinued before receiving treatment due to a protocol violation) | 12
Completed | 0 | 0
Not Completed | 10 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 4 | 6
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorinostat Once Daily Dose Schedule | Vorinostat Thrice Daily Dose Schedule | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.0 (18.5) | 64.0 (10.5) | 66.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  White | 9 | 10 | 19
  Black | 0 | 1 | 1
  Asian | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Scale Status [Number; unit: participants] — ECOG Scale: 0 = Normal Activity, 1 = Symptoms, but ambulatory, 2 = In bed <50% of the time, 3 = In bed >50% of the time, 4 = 100% Bedridden, 5 = Dead
  participants
    0 = Normal Activity | 4 | 10 | 14
    1 = Symptoms, but ambulatory | 4 | 1 | 5
    2 = In bed < 50% of the time | 1 | 1 | 2
International Prognostic Scoring System Risk (IPSS) [Number; unit: Participants] — IPSS Risk: Low [Score = 0; Time to Acute myeloid leukemia (AML) (yrs) = 9.4; Median Survival (yrs) = 5.7]
  IPSS Risk: INT-1 [Score = 0.5 - 1; Time to AML (yrs) = 3.3; Median Survival (yrs) = 3.5]
  IPSS Risk: INT-2 [Score = 1.5 - 2; Time to AML (yrs) = 1.1; Median Survival (yrs) = 1.2]
  IPSS Risk: High [Score = >2; Time to AML (yrs) = 0.2; Median Survival (yrs) = 0.4]
  Participants
    Low | 3 | 4 | 7
    Intermediate-1 | 6 | 8 | 14
Prior Myelodysplastic Syndromes Therapy [Number; unit: Participants]
  Yes | 6 | 3 | 9
  No | 3 | 9 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders and Number of Non-responders Defined by International Working Group Response Criteria
Description: Number of responders is defined as the number of patients in the analysis population who have complete response (CR), partial response (PR), or hematologic improvement (HI) per International Working Group Response Criteria during the course of the study. Confirmation of CR or PR will require a second assessment performed 4 weeks or more after the initial assessment. Confirmation of HI will require a second assessment performed 8 weeks or more after the initial assessment. Number of non-responders is defined as the number of patients who did not achieve CR, PR or HI in the study.
Time Frame: 2 Years
Population: Full analysis set (FAS) population is the analysis population. This population consists of all randomized patients who have received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Vorinostat Once Daily Dose Schedule | Vorinostat Thrice Daily Dose Schedule
Number analyzed (Participants) | 9 | 12
Participants
  Responder | 0 | 0
  Non-responder | 9 | 12

2. Primary Outcome: Safety and Tolerability as Assessed by the Number of Participants With Adverse Events.
Time Frame: Every 21 days while on therapy and at 30 days after the last dose of study therapy
Measure: Number; unit: Participants
Arm/Group | Vorinostat Once Daily Dose Schedule | Vorinostat Thrice Daily Dose Schedule
Number analyzed (Participants) | 9 | 12
Participants
  With one or more adverse events | 9 | 12
  With no adverse events | 0 | 0
  With drug-related adverse events | 4 | 11
  With serious adverse events | 2 | 5
  With serious drug-related adverse events | 0 | 2

ADVERSE EVENTS:
Time Frame: Serious and non-serious adverse experiences occurring from the time of consent up through 30 days after the last dose of study drug were reported.
Description: One patient was randomized to the Once Daily Dose Schedule, but discontinued before receiving study medication due to a protocol violation and is not included in the safety assessment.
Arm/Group | Vorinostat Once Daily Dose Schedule | Vorinostat Thrice Daily Dose Schedule
Serious Adverse Events (participants affected / at risk) | 2/9 | 5/12
Other Adverse Events (participants affected / at risk) | 9/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat Once Daily Dose Schedule (N=9) | Vorinostat Thrice Daily Dose Schedule (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Eye infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorinostat Once Daily Dose Schedule (N=9) | Vorinostat Thrice Daily Dose Schedule (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye irritation (Eye disorders) | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 11
Dry mouth (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 9
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Tongue discolouration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 5
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 4 | 7
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0
Haematocrit decreased (Investigations) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Balance disorder (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3
Dysgeusia (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This trial was terminated because the pre-specified futility criterion was met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.